CLINICAL TRIAL: NCT05700591
Title: A Phase III Trial to Assess the Efficacy and Safety of Recombinant Human Prourokinase in the Treatment of Acute Acute Ischaemic Stroke in 4.5 Hours After Stroke Onset
Brief Title: rhPro-UK in Acute Ischaemic Stroke Within 4.5 Hours of Stroke Onset Trial 2(PROST-2)
Acronym: PROST-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASLY-B1440-CTP-Ⅲc
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhPro-UK (Experimental): Recombinant Human Pro-urokinase (rhPro-UK)
  Interventions: Drug: rhPro-UK
- rt-PA (Active Comparator): Alteplase(rt-PA)
  Interventions: Drug: rt-PA

INTERVENTIONS:
Drug: rhPro-UK — 35 mg, administered intravenously with a bolus of 15 mg within 3 minutes and the remainder by continuous infusion within 30 minutes
  Arms: rhPro-UK
Drug: rt-PA — 0.9 mg/kg (maximum 90 mg), with 10% administered intravenously as a bolus, followed by 90% infusion within 1 hour
  Arms: rt-PA

SUMMARY:
Intravenous thrombolysis is the first-line therapy in patients with acute ischemic stroke within 4·5 hours of symptom onset, and recombinant tissue plasminogen activator (alteplase) is the preferred thrombolytic agent for this purpose.

RhPro-UK is a specific plasminogen activator. rhPro-UK only acts on occlusive thrombus and has little effect on hemostatic thrombus. In addition, rhPro-UK does not form covalent complexes with protease inhibitors in plasma, so the concentrations of rhpro-UK and protease inhibitors in the blood do not decrease compared with alteplase. Therefore, rhPro-UK therapies have a potential advantage of less systemic bleeding in treated subjects. Data from several previous studies suggest that rhPro-UK is efficacious when used to treat patients with acute myocardial infarction. On April 2, 2011, rhPro-UK injection was approved by the National Medical Products Administration to treat acute myocardial infarction. Since then, rhPro-UK has been widely used to treat myocardial infarction in China.

Since 2016, a phase 2 clinical trial was carried to explore the dosing of rhPro-UK in patients with acute ischemic stroke, followed by another study with a sample size of 680 patients to initially validate the efficacy and safety of the proposed dose of 35mg. The results of these studies suggested that rhPro-UK was effective, and there were no safety concerns. To further prove the efficacy and safety of rhPro-UK in patients with acute ischemic stroke, investigators conducted this phase 3 study (PROST-2).

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed as acute ischemic stroke (according to the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018).
2. 18 years or older, male or female.
3. NIH Stroke Scale（NIHSS）scores of 4 to 25.
4. Treatment within 4.5 hours after stroke onset.
5. The symptoms of stroke last at least 30 minutes without significant improvement before treatment.
6. Informed consent by patient or by patient's guardians.

Exclusion Criteria:

1. Prestroke modified rankin scale of ≥2.
2. Large areas of hypodense ischaemic changes on baseline CT（Infarction area> 1/3 of the middle cerebral artery feeding area）.
3. Intracranial hemorrhage.
4. Previous history of intracranial hemorrhage.
5. Severe cerebral trauma or stroke history within 3 months.
6. Intracranial tumor or giant intracranial aneurysm.
7. Intracranial or intraspinal surgery within the past 3 months.
8. Gastrointestinal or urinary bleeding within the past 3 weeks.
9. History of major surgical procedures or severe trauma within the last 2 weeks (investigator evaluation).
10. Puncture in 1 week which can not be oppressed.
11. Active visceral hemorrhage.
12. Aortic arch dissection.
13. Bacterial endocarditis or pericarditis.
14. Planned for thrombectomy.
15. Patients with systolic blood pressure ≥ 185 mmHg or diastolic blood pressure ≥ 110 mmHg after anti-hypertension treatment.
16. High risk of acute hemorrhage include platelet count<10^9/L.
17. Received low molecular weight heparin or heparin within 24 hours.
18. Using of thrombin inhibitors or factor Xa inhibitor within the past 48 hours.
19. Using of oral anticoagulant drugs and PT >15s or INR >1.7.
20. Patients with epilepsy or other mental disorders that could not be adhered to at the beginning of stroke.
21. Blood glucose < 2.8 mmol/L or > 22.2 mmol/L.
22. Allergies to rhPro-UK or rt-PA active ingredients or other components.
23. Pregnant women or beastfeeding women.
24. Participants in other clinical trials within the past month.
25. The investigator believes that the patient is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1552 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with excellent functional outcome at 90 days | 90±7 days
  A score of 0 or 1 on the modified Rankin scale(which ranges from 0 [no symptoms] to 6 [death]) at 90 days indicated an excellent functional outcome.

SECONDARY OUTCOMES:
The proportion of patients with independent functional outcome at 90 days | 90±7 days
  A score of 0-2 on the modified Rankin scale(which ranges from 0 [no symptoms] to 6 [death]) at 90 days indicated an independent functional outcome.
Functional handicap | 90±7 days
  The distribution of the modified Rankin scale(which ranges from 0 [no symptoms] to 6 [death]) at 90 days
The proportion of patients with neurological improvement at 24 hours | 22-36 hours
  A reduction in NIHSS score of ≥4 or a score of 0-1 indicated neurological improvement. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
The proportion of patients with neurological improvement at 7 days | 7 ±2 days
  A reduction in NIHSS score of ≥4 or a score of 0-1 indicated neurological improvement. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
The change of neurological function at 24 hours | 22-36 hours
  NIHSS score was used to assess neurological function. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
The change of neurological function at 7 days | 7 ±2 days
  NIHSS score was used to assess neurological function. Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe cerebral infarcts.
Self-care ability in daily life | 90±7 days
  The Barthel Index(which ranges from 0[complete dependence on help with activities of daily living] to 100[independence]) of 95-100 at 90 days
All-cause death within 7 days | 7 days
All-cause death within 90 days | 90 days
Symptomatic intracranial hemorrhage defined as SITS-MOST | 22-36 hours
Symptomatic intracranial hemorrhage defined as ECASSIII | 7 days
Any intracranial hemorrhage | 7 days
Any systematic bleeding event（defined as ISTH） | 7 days

CONTACTS AND LOCATIONS:
Locations (72):
- China (72):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Huizhou First Hospital, Guangdong, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Handan Central Hospital, Handan, Hebei
  - Hengshui People's Hospital (Harrison International Peace Hospital), Hengshui, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - General Hospital of Pingmei Shenma Medical Group, Pingdingshan, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Tongji Hospital affiliated to Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Baogang Hospital of Inner Mongolia, Baotou, Inner Mongolia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science & Technology, Baotou, Inner Mongolia
  - Keshiketeng Hospital of Traditional Chinese Medicine and Mongolian Medicine, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - General Hospital of Xuzhou Coal Mining Group, Xuzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Guowen Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Jilin Neuropsychiatric Hospital, Siping, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Ansteel Group General Hospital, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - Beipiao Central Hospital, Chaoyang, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Fukuang General Hospital of Liaoning Health Industry Group, Fushun, Liaoning
  - Fuxinkuang General Hospital of Liaoning Health Industry Group, Fuxin, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The PLA General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Xianyang Hospital Of Yan'an University, Xianyang, Shaanxi
  - Dezhou People's Hospital, Dezhou, Shandong
  - Tengzhou Central People's Hospital, Dezhou, Shandong
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Jinan City People's Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - First People's Hospital of Tancheng, Tancheng, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - Zhejiang Taizhou Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Gu HQ, Feng B, Li H, Wang X, Dong Q, Fan D, Xu Y, Zhu S, Dai H, Wei Y, Wang Z, Lu G, Ma Y, Li Z, Wang Y, Meng X, Zhao X, Liu L, Wang Y; PROST-2 investigators. Safety and efficacy of intravenous recombinant human prourokinase for acute ischaemic stroke within 4.5 h after stroke onset (PROST-2): a phase 3, open-label, non-inferiority, randomised controlled trial. Lancet Neurol. 2025 Jan;24(1):33-41. doi: 10.1016/S1474-4422(24)00436-8. Epub 2024 Nov 29. PMID 39617030
- [Derived] Li S, Gu HQ, Feng B, Dong Q, Fan D, Xu Y, Zhu S, Wang Y. RhPro-UK in acute ischemic stroke within 4.5 h of stroke onset trial-2 (the PROST-2 study): Rationale and design of a multicenter, prospective, randomized, open-label, blinded-endpoint, controlled phase 3 non-inferiority trial. Int J Stroke. 2024 Dec;19(10):1182-1187. doi: 10.1177/17474930241265654. Epub 2024 Aug 3. PMID 38907679